CLINICAL TRIAL: NCT04477044
Title: Use of Point-of-View Camera to Faciliate Learning of Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, NUS Anaesthesia, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NUS IRB B-15-274
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Intubation; Difficult or Failed; Anesthesia
Keywords: Medical Education; Intubation

STUDY DESIGN:
Intervention Model Description: The participants will be randomised to 2 groups, either in the study group having a GoPro Hero4 camera mounted on their head or control group with no GoPro Hero4 camera mounted on their head
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No GoPro (No Intervention): No GoPro Hero4 to be mounted on the participant's head while he/she performs intubation on a manikin.
- GoPro (Experimental): GoPro Hero4 to be mounted on the participant's head while he/she performs intubation on a manikin.
  Interventions: Other: Study Group

INTERVENTIONS:
Other: Study Group — GoPro Hero4 to be mounted on the participant's forehead while performing intubation on a manikin.
  Other Names: GoPro
  Arms: GoPro

SUMMARY:
The study team proposes that mounting a point-of-view camera on the student's head will enable the team to view what the student is seeing in real-time when intubating with a normal laryngoscope. This will allow the team to guide the students accurately. When used in conjunction with the established simulation programme in the department, it is believed that this will improve the learning and retention of this skill when compared to standard teaching.

DETAILED DESCRIPTION:
The ability to correctly perform an endotracheal intubation is a life-saving skill that every doctor should possess. It is an integral part of established protocols for resuscitation and advanced cardiac life support (ACLS). It is an essential procedural skill that is taught to all students at the Yong Loo Lin School of Medicine, NUS. It is also recommended by the American Association of Medical Colleges as an essential procedural skill for medical students to learn.

Timely and correctly performed endotracheal intubation can be life-saving because it maintains and protects the airway, reliably provides adequate tidal volumes, frees the hands of rescuers, allows the removal of airway secretions and provides a route for giving drugs. However, poorly performed endotracheal intubation exposes patients to the life-threatening risks associated with the unrecognised misplacement of a tracheal tube and leads to delays in resuscitative efforts.

Unfortunately, there is a comparatively high failure rate associated with endotracheal intubation because this skill is difficult to learn and retain. Mulcaster et al reported that, to achieve a 90% intubation success rate, a mean of 47 intubation attempts were required. In a similar study, Konrad et al found that a mean of 57 attempts were required to achieve a 90% intubation success rate. This difficulty in learning is compounded by the finding that, without repeated practice, the ability to perform endotracheal intubation successfully diminishes rapidly. The intubation success rate of infrequent users who have successfully learned to intubate has been shown to fall to as little as 57% after only 6 months. Clearly, there is a need to improve the learning and retention of endotracheal intubation.

The PI previously published a randomized controlled trial in the journal Medical Education to study the utility of experiential learning on a simulator in the learning and retention of this skill. It was showed that with experiential learning, more students were able to intubate a manikin at 3 months (64.5% vs. 36.9%, p<0.001). With repeated learning (refresher every 3 months), 86% of students were able to successfully perform endotracheal intubation at 12 months.

However, there are limitations to acquiring this skill on a simulator, as it has been argued that expertise gained on manikins may not translate into successful intubations in patients. Learning on actual patients is desirable, but impractical given the large number of students in our medical school. On average, each YLLSoM student only intubates between 3-5 patients, far less than the 47-57 endotracheal intubations necessary to gain expertise as cited earlier. Combining the learning experiences on the simulator with that on actual patients appears to be the best solution.

Therefore it is important to optimize the limited learning opportunities on patients. However, this is often difficult because the mouth is small, and the view of the pharyngeal structures is limited. The tutor will not be able to view what the student is seeing as there is only one line of vision. More recently, video-laryngoscopes, which are laryngoscopes with a camera at its tip, have emerged as an effective means of teaching endotracheal intubation. However, the technique of using the video-laryngoscope differs from using the common laryngoscope due to its different shape and the requirement that the student looks at the screen rather than into the patient's mouth. Hence it is unclear if the ability to successfully perform endotracheal intubation with a video-laryngoscope necessarily translates into the ability to perform endotracheal intubation with a normal laryngoscope.

The study team proposes that mounting a point-of-view camera on the student's head will enable the team to view what the student is seeing in real-time when intubating with a normal laryngoscope. This will allow the team to guide the students accurately. When used in conjunction with the established simulation programme in the department, it is believed that this will improve the learning and retention of this skill when compared to standard teaching.

Methods:

Students will be randomised into 2 groups. For the study group, students will have a GoPro Hero4 camera mounted on their head which will be linked via Wi-Fi to allow real-time streaming of the view onto a laptop, while students in control group will have a regular type of tutorial and practicing session. Data such as time to successful intubation and Cormack Lehane laryngoscopy view will be recorded. At the end of the session, tutors will use a debrief guide to give feedback to students. Students from the study group will be given a questionnaire to be completed at the end of the session.

These students will be recalled 3 months later. Each student will individually be assessed on his or her intubation skill using 2 different manikin: a normal airway manikin and a difficult airway manikin. All the students will be wearing the GoPro Hero4 this time round. Data such as time to successful intubation and Cormack Lehane laryngoscopy view will be recorded. Students will be given feedback as appropriate by tutors for their learning purposes using the same debrief guide. There will be questionnaires for both students and tutors to fill in this time.

ELIGIBILITY:
Inclusion Criteria:

* All medical students rotating through a 2-week posting in Anaesthesia at NUHS during Year 4 of medical school

Exclusion Criteria:

* NIL

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Intubation Timing between GoPro and non-GoPro group at first intubation session | During procedure of first intubation session
  To record the difference in time taken for successful intubation of the manikin between the GoPro and non-GoPro group
Intubation Timing between GoPro and non-GoPro group at 3 months follow-up session | During procedure of 3-month follow-up session
  To record the difference in time taken for successful intubation of the manikin between the GoPro and non-GoPro group

SECONDARY OUTCOMES:
Usefulness of GoPro in learning | Immediately after first intubation tryout session and follow-up session 3 months later
  To find out the usefulness of GoPro in learning using a questionnaire comprising of yes/no questions

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, Principal Investigator — National University of Singapore
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulcaster JT, Mills J, Hung OR, MacQuarrie K, Law JA, Pytka S, Imrie D, Field C. Laryngoscopic intubation: learning and performance. Anesthesiology. 2003 Jan;98(1):23-7. doi: 10.1097/00000542-200301000-00007. PMID 12502974
- [Background] Konrad C, Schupfer G, Wietlisbach M, Gerber H. Learning manual skills in anesthesiology: Is there a recommended number of cases for anesthetic procedures? Anesth Analg. 1998 Mar;86(3):635-9. doi: 10.1097/00000539-199803000-00037. PMID 9495429
- [Background] Ti LK, Chen FG, Tan GM, Tan WT, Tan JM, Shen L, Goy RW. Experiential learning improves the learning and retention of endotracheal intubation. Med Educ. 2009 Jul;43(7):654-60. doi: 10.1111/j.1365-2923.2009.03399.x. PMID 19573188